CLINICAL TRIAL: NCT00430885
Title: Phase III Study of Intravenous Immunglobulin (IVIG) in Patients With Heart Failure After Myocardial Infarction
Brief Title: Effect of Intravenous Immunglobulin (IVIG) After Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Lars Gullestad, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 175464/V50; NFR 175464/V50
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Heart failure; Myocardial infarction; Patients with acute myocardial infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction | interventions — Octagam; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: Octagam (IVIG)
- Octagam (IVIG) (Experimental): Octagam (IVIg) is intravenous immunglobulin
  Interventions: Drug: Octagam (IVIG)

INTERVENTIONS:
Drug: Octagam (IVIG) — Intravenous immunoglobulin 0.4 g/kg given as infusion
  Other Names: Intravenous immunoglobulin 0.4 g/kg given as infusion

SUMMARY:
The instigators hypothesize that IVIG, given in the acute phase following MI in patients at risk for developing HF, will improve cardiac performance, and by attenuating cardiac remodeling in this phase, such therapy will prevent the development of chronic HF resulting in long term beneficial effect also after the therapy has been stopped.

DETAILED DESCRIPTION:
This double-blind placebo-controlled study represents a new approach to cardiovascular disease. The project deals with unresolved issues in the intersection between cardiology, immunology and molecular biology.

IVIG/placebo will be given as an induction therapy for 5 days and thereafter as monthly infusions for 5 months. Change in left ventricular remodeling will be assessed at baseline, and 6 and 12 months with MRI and echocardiography.

The objectives are:

1. The primary objective of this study is to evaluate the effect on IVIG on LV remodeling and function: LV remodeling will be evaluated with magnetic resonance imaging (MRI) which offers an unsurpassed precision in the measurements of heart volumes and function. End points will be LV-end systolic and diastolic volume (LVESV, LVEDV), regional wall motion score index (WMSI), and LV-ejection fraction (LV-EF).
2. The secondary objective of this study is to evaluate the effect on IVIG on the myocardial marker B-Type Natriuretic Peptide (BNP). BNP is a sensitive marker of the degree of HF besides being a prognostic indicator 18-20.
3. The tertiary objective of this study is to evaluate the effect on IVIG on:

   a. Quality of life. b. Effect on New York Heart Association (NYHA) functional class. c. Effect on immunological variables. i. Inflammatory cytokines such as TNF-alpha, IL-6, IL-18. ii. Anti-inflammatory cytokines such as IL-10 and transforming growth factor beta iii. Chemokines such as monocyte chemoattractant protein 1, IL-8 and CCL21. iv. Regulators of hypertrophy such as matrix metalloproteinases, their endogenous inhibitors (i.e., TIMPs) and procollagen III N-terminal.

   d. Effect on neurohormones. e. Withdrawals. f. Side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-80 years
* Have a recent MI (<5days)
* Have ASAT >100 U/L or CKMB > 50 U/L.
* Have LVEF <40%.
* Are on optimal medical treatment and considered unsuitable for surgical intervention.

Exclusion Criteria:

* Evidence of unstable disease, concomitant ischemia or unstable angina during the hospitalization.
* Significant concomitant disease such as infections, pulmonary disease or connective tissue disease.
* Participating in other studies.
* Inability to participate.
* Diseases that require surgery.
* Planned revascularisation.
* Known hypersensitivity to IVIG.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
1. The effect on IVIG on LV remodeling (volume and ejection fraction) and function as assessed by MRI | 2009

SECONDARY OUTCOMES:
2. Effect on IVIG on B-Type Natriuretic Peptide (BNP). | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD, PhD, Principal Investigator
Locations (1):
- Rikshospitalet University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Gullestad L, Orn S, Dickstein K, Eek C, Edvardsen T, Aakhus S, Askevold ET, Michelsen A, Bendz B, Skardal R, Smith HJ, Yndestad A, Ueland T, Aukrust P. Intravenous immunoglobulin does not reduce left ventricular remodeling in patients with myocardial dysfunction during hospitalization after acute myocardial infarction. Int J Cardiol. 2013 Sep 20;168(1):212-8. doi: 10.1016/j.ijcard.2012.09.092. Epub 2012 Oct 6. PMID 23046599